CLINICAL TRIAL: NCT00097097
Title: Neonatal Resuscitation in Zambia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GN 03; U01HD043464 (NIH)
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Asphyxia Neonatorum; Neonatal Mortality; Hypoxic Ischemic Encephalopathy
Keywords: Asphyxia; Neonatal mortality; Neonatal morbidity; Hypoxic ischemic encephalopathy; Neurodevelopmental impairment; Neonatal resuscitation; Global Network; Zambia; Africa; Cerebral palsy; Child health; International
MeSH Terms: conditions — Asphyxia Neonatorum; Hypoxia-Ischemia, Brain; Asphyxia; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Neonatal Resuscitation

SUMMARY:
Asphyxia is a leading cause of neonatal death in Zambia. This study will be conducted in two cities in Zambia to determine if the combined Neonatal Resuscitation Program/Essential Newborn Care Program compared to the new World Health Organization (W.H.O.) basic perinatal care education of health care providers (Essential Newborn Care Program) results in reduced mortality due to perinatal asphyxia.

DETAILED DESCRIPTION:
Birth asphyxia (defined as "failure to initiate and sustain breathing at birth") has been identified by the World Health Organization (WHO) as the most frequent cause of early deaths worldwide, accounting for about 20% of neonatal mortality. Although prompt resuscitation after birth can prevent many of the deaths and reduce disabilities in survivors from birth asphyxia, the WHO has concluded that resuscitation is often not initiated or the methods used are inadequate or wrong. The Neonatal Resuscitation Program (NRP) has been universally accepted in the developed world but has had limited dissemination in many developing countries, including Zambia. The primary hypothesis of this study is that implementation of the combined Neonatal Resuscitation Program/WHO Essential Newborn Care (ENC) Program, compared to basic neonatal care education of health care providers (ENC only) will result in reduced neonatal 7-day mortality. This trial will be performed in two Zambian cities: Lusaka and Ndola. Training in data collection will be conducted in order to establish baseline data on mortality and asphyxia. Following this time period, all centers will receive the ENC training and continue to collect data for 7 months. The clinics will then receive NRP Training and collect data for a 12-month period.

The primary outcome will be a decrease in neonatal 7-day mortality following the NRP training when compared to the ENC-only time period. Secondary outcomes will include neonatal mortality due to perinatal asphyxia, mortality or hypoxic ischemic encephalopathy (HIE) at 7 days, need for advanced resuscitation, Apgar scores at 5 minutes, sustainability of the program, as well as providers' self efficacy, competence, and performance in neonatal resuscitation.

ELIGIBILITY:
Inclusion criteria:

* Live birth infants with birth weight ≥ 1500 g
* Infants who are born at participating health centers in Lusaka and Ndola, Zambia
* No lethal malformations

Exclusion criteria:

* Stillbirths
* Infants with suspected/confirmed lethal malformations (e.g. anencephaly, Trisomy 13 or 18, or cyanotic or left sided congenital heart disease that will not be repaired)
* Any infant who is transported/brought to the center after delivery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40000
Dates: Start 2004-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality at 7 days

SECONDARY OUTCOMES:
Neonatal mortality due to perinatal asphyxia
Self efficacy, knowledge, performance, and competence in neonatal resuscitation
Apgar scores at 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Elwyn Chomba, MBChB, DCH, MRCP, Principal Investigator — University Teaching Hospital, Lusaka, Zambia
Locations (1):
- University of Zambia, Lusaka, Zambia

REFERENCES:
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org